CLINICAL TRIAL: NCT00130663
Title: Recognition of Abnormal Pediatric Blood Pressures in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 219405; 219405
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2007-10-22 (Estimated); Status verified 2007-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Device: PDA blood pressure screening program and chart reminder

SUMMARY:
This study will look at general pediatricians' effectiveness at screening children for elevated blood pressure values in the primary care setting. Two new screening tools will be introduced and their effectiveness will be measured against current practice by way of medical chart review.

ELIGIBILITY:
Inclusion Criteria:

* Health care supervision visit
* Documented measured blood pressure and height
* Between the ages of 3 years and 17 years

Exclusion Criteria:

* Younger than 3 years of age
* Older than 17 years of age
* No documented blood pressure measurement
* Not a health supervision encounter

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2006-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
written documentation by MD in medical record acknowledging elevated BP

SECONDARY OUTCOMES:
compliance with interventions

CONTACTS AND LOCATIONS:
Overall Officials: Douglas J McLaughlin, MD, Principal Investigator — Pediatric Academic Association/Ohio State University School of Medicine